CLINICAL TRIAL: NCT00064337
Title: S0115, A Phase II Trial Evaluating Modified High Dose Melphalan (100 mg/m) And Autologous Peripheral Blood Stem Cell Supported Transplant (SCT) For High Risk Patients With Multiple Myeloma And/Or Light Chain Amyloidosis (AL Amyloidosis) (A BMT Study)
Brief Title: S0115, High-Dose Melphalan and Autologous Peripheral Stem Cell Transplantation in Treating Patients With Multiple Myeloma or Primary Systemic Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0115; S0115 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Multiple Myeloma; Plasma Cell Myeloma
Keywords: primary systemic amyloidosis; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis | interventions — Filgrastim; Cyclophosphamide; Dexamethasone; Melphalan; Thalidomide; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): MM Induction: dexamethasone 20mg/d PO Days 1-4, 9-12 and 17-20 every 35 days for 2 cycles and thalidomide 200 mg/d PO Days 1-70.
  Mobilization and SC Collection:
  MM, MM+AL, MM+LCD: cyclophosphamide 2.5 gm/m2 IV Day 1; mesna 800 mg/m2 IV Day 1 x 3 doses; G-CSF 10 mcg/kg/d SQ Day 2 through day prior to last leukapheresis.
  Amyloid or LCDD-Only: G-CSF 16 mcg/kg/d SQ Days 1-3 (continued daily until the day prior to the last day of stem cell collection).
  Conditioning/Transplant - Modified HighDose Melphalan (given for both transplants): melphalan 100 mg/m2/d IV over 20 mins Day -2; PBSC infusion >/= 3.5 x 10^6 CD34+ cells/kg IV Day 0.
  Maintenance (MM only): dexamethasone 40 mg/d PO Days 1-4 every 28 days and thalidomide 100 mg/d PO daily - given for one year, followed by dexamethasone 40 mg/d PO Days 1-4 every 28 days and thalidomide 100 mg/d PO daily - given for one year.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: dexamethasone; Drug: melphalan; Drug: thalidomide; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: dexamethasone
Drug: melphalan
Drug: thalidomide
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as melphalan work in different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with donor peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving melphalan together with autologous stem cell transplantation works in treating patients with multiple myeloma or primary systemic amyloidosis.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine overall survival of patients with high-risk multiple myeloma, primary systemic amyloidosis, or light chain deposition disease treated with two courses of modified high-dose melphalan and autologous peripheral blood stem cell transplantation.
* Determine the hematologic response in patients treated with this regimen.
* Determine the qualitative and quantitative toxic effects of this regimen in these patients.
* Determine the prognostic significance of cytogenetic markers in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to disease (high-risk multiple myeloma vs primary systemic amyloidosis vs both).

* Induction therapy (multiple myeloma patients only): Patients receive oral dexamethasone on days 1-4, 9-12, and 17-20 and oral thalidomide daily on days 1-35. Treatment repeats every 35 days for 2 courses in the absence of disease progression or unacceptable toxicity.
* Mobilization and stem cell collection:

  * Multiple myeloma patients: Within 28-35 days after completion of induction therapy, patients receive cyclophosphamide IV over 2-3 hours on day 1 and filgrastim (G-CSF) subcutaneously (SC) daily beginning on day 2 and continuing through the day before the last leukapheresis. Usage of mesna IV on day 1 (prior to and twice after cyclophosphamide administration is recommended).
  * Primary systemic amyloidosis patients: Patients receive G-CSF SC daily beginning on day 1 and continuing through the day before the last leukapheresis.

All patients undergo leukapheresis for the collection of stem cells until the target number of CD34+ cells is reached.

* Conditioning regimen: Within 1-4 weeks after mobilization, patients receive modified high-dose melphalan IV over 20 minutes on day -2.
* Peripheral blood stem cell (PBSC) reinfusion: PBSCs are reinfused on day 0. Patients receive G-CSF SC daily beginning on day 1 and continuing until blood counts recover.

Patients undergo a second autologous PBSC transplantation within 3-6 months, but no later than 12 months, after the first transplantation.

* Second conditioning regimen: Patients receive modified high-dose melphalan IV over 20 minutes on day -2.
* Second PBSC infusion: PBSCs are infused on day 0.
* Maintenance regimen (multiple myeloma patients only): Between 4-8 weeks after the second transplantation, patients with no progressive disease receive oral dexamethasone once daily on days 1-4 and oral thalidomide once daily on days 1-28. Courses repeat every 28 days for 2 years in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3 and 6 months and then annually thereafter.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 20-25 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* At least 1 of the following diagnoses:

  * Multiple myeloma

    * Stage II or III disease
    * At least 1 of the following must be present:

      * Serum M-protein of IgG, IgA, IgD, IgE greater than 1.0 g/dL
      * Urinary M-protein (Bence-Jones) at least 200 mg/24 hours
    * No IgM peaks except in patients who have physiologic criteria to support a diagnosis of multiple myeloma (e.g., bony lesions, myeloma kidney-cast nephropathy, absence of adenopathy [unless pathology-proven to be plasma cell infiltration])
    * No monoclonal gammopathy of undetermined significance
    * No indolent or smoldering myeloma
    * No disease progression on prior thalidomide or dexamethasone
  * Histologically confirmed primary systemic amyloidosis

    * No senile, secondary, localized, dialysis-related, or familial amyloidosis
    * No severe cardiac involvement

      * No pre-exertional syncope, ventricular arrhythmia, or symptomatic pleural effusions associated with cardiac involvement
  * Light Chain Deposition Disease alone or in combination with multiple myeloma meeting the following criteria:

    * Deposition of granular material containing free light chains/immunoglobulins that did not bind Congo red
    * Evidence of plasma cell dyscrasia (i.e., monoclonal gammopathy in the serum or urine by immunofixation electrophoresis and/or clonal plasmacytosis) on bone marrow biopsy by immunohistochemistry and/or elevated serum-free light chain concentration
* Must have been diagnosed within the past year
* Concurrent enrollment in the myeloma repository protocol SWOG-S0309 must be offered

PATIENT CHARACTERISTICS:

Age

* 18 and over (patients with amyloidosis only OR patients with amyloidosis and multiple myeloma OR patients with multiple myeloma only with poor renal function) OR
* 70 and over (patients with multiple myeloma only with or without poor renal function)

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2.5 times upper limit of normal (ULN)
* SGOT or SGPT no greater than 2.5 times ULN

Renal

* No hemodialysis within 2 hours of melphalan or stem cell infusion

Cardiovascular

* See Disease Characteristics
* Hemodynamically stable (i.e., systolic blood pressure > 90 mm Hg in a lying position within the past 42 days)
* No myocardial infarction within the past 6 months
* No congestive heart failure
* No arrhythmia refractory to medical therapy
* LVEF greater than 45% by echocardiogram or MUGA

Pulmonary

* See Disease Characteristics
* No history of chronic obstructive or chronic restrictive pulmonary disease
* Pulmonary function studies (e.g., FEV_1 and FVC) at least 50% of predicted
* DLCO at least 50% of predicted
* Normal high resolution CT scan of the chest and acceptable arterial blood gases (i.e., PO_2 greater than 70) required for patients unable to complete pulmonary function tests due to bone pain or fracture

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

  * Multiple myeloma patients receiving thalidomide must use 2 methods of effective contraception for at least 4 weeks before, during, and for at least 4 weeks after discontinuation of thalidomide
* HIV negative
* No other concurrent significant medical condition
* No concurrent uncontrolled life-threatening infection
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics
* Prior cumulative melphalan dose no more than 200 mg
* No other concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent hormonal therapy

Radiotherapy

* No concurrent radiotherapy

Surgery

* Not specified

Other

* Recovered from prior therapy
* Prior or concurrent bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2004-01; Primary Completion 2012-05 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaishali Sanchorawala, MD, Study Chair — Boston Medical Center; David C. Seldin, MD, PhD, Study Chair — Boston Medical Center
Locations (35):
- United States (35):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California Davis Cancer Center, Sacramento, California
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Northwest Cancer Specialists at Rose Quarter Cancer Center, Portland, Oregon
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: MM Induction: dexamethasone 20mg/d PO Days 1-4, 9-12 and 17-20 every 35 days for 2 cycles and thalidomide 200 mg/d PO Days 1-70.
  Mobilization and SC Collection: MM, MM+AL, MM+LCD: cyclophosphamide 2.5 gm/m2 IV Day 1; mesna 800 mg/m2 IV Day 1 x 3 doses; G-CSF 10 mcg/kg/d SQ Day 2 through day prior to last leukapheresis.
  Amyloid or LCDD-Only: G-CSF 16 mcg/kg/d SQ Days 1-3 (continued daily until the day prior to the last day of stem cell collection).
  Conditioning/Transplant - Modified HighDose Melphalan (given for both transplants): melphalan 100 mg/m2/d IV over 20 mins Day -2; PBSC infusion >/= 3.5 x 10^6 CD34+ cells/kg IV Day 0.
  Maintenance (MM only): dexamethasone 40 mg/d PO Days 1-4 every 28 days and thalidomide 100 mg/d PO daily - given for one year, followed by dexamethasone 40 mg/d PO Days 1-4 every 28 days and thalidomide 100 mg/d PO daily - given for one year.
  filgrastim
  cyclophosphamide
  dexamethasone
  melphalan
  thalidomide
  peripheral blood
Period: PBSCC or Induction/PBSCC
Arm/Group | Treatment
Started | 93 (104 patients were registered, 93 of whom were eligible and analyzable.)
Completed | 73
Not Completed | 20
Not completed — Not protocol-specified | 7
Not completed — Adverse Event | 6
Not completed — Progression | 3
Not completed — Patient Refusal | 2
Not completed — Death | 2
Period: Transplant
Arm/Group | Treatment
Started | 67 (6 patients who completed PBSCC or Induction/PBSCC did not begin Transplant)
Completed | 46
Not Completed | 21
Not completed — Adverse Event | 9
Not completed — Not protocol-specified | 5
Not completed — Death | 3
Not completed — Patient Refusal | 2
Not completed — Progression | 2
Period: Maintenance
Arm/Group | Treatment
Started | 13 (Only patients with High Risk MM or AL + MM were allowed to enroll to Maintenance treatment.)
Completed | 3
Not Completed | 10
Not completed — Adverse Event | 3
Not completed — Progression | 2
Not completed — On treatment at time of analysis | 2
Not completed — Not protocol-specified | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 93
Age, Continuous [Median (Full Range); unit: years] | 65 [33 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 58

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Time from initial registration until death or date of last contact, whichever occurs first, for up to 5 years from the date of the last patient registration.
Time Frame: 5 years from initial registration, or until death, whichever occurred earlier, on average, about 4.5 years
Population: Eligible and analyzable patients only.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment
Number analyzed (Participants) | 93
Months | 68 [42 to NA] — The upper limit of the 95% CI for the median had not yet been reached at time of analysis.

2. Secondary Outcome: Hematologic Response
Time Frame: Until off study
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 23
Participants | 8

ADVERSE EVENTS:
Groups:
- PBSCC or Induction/PBSCC: Induction/PBSCC - High Risk MM or MM with Light Chain Amyloidosis/Light Chain Disposition; PBSCC - Light Chain Amyloidosis/Light Chain Disposition
- Autologous Transplants: Autologous Transplants � All patients
- Dex/Thal: Dex/Thal - High Risk MM or MM with Light Chain Amyloidosis/Light Chain Disposition
Arm/Group | PBSCC or Induction/PBSCC | Autologous Transplants | Dex/Thal
Serious Adverse Events (participants affected / at risk) | 4/92 | 3/65 | 1/12
Other Adverse Events (participants affected / at risk) | 83/92 | 62/65 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PBSCC or Induction/PBSCC (N=92) | Autologous Transplants (N=65) | Dex/Thal (N=12)
Cardiac General-Other (Cardiac disorders) | 1 | 0 | 0
Cardiac-ischemia/infarction (Cardiac disorders) | 0 | 1 | 0
Left ventricular diastolic dysfunction (Cardiac disorders) | 1 | 0 | 0
SVT and nodal arrhythmia - Nodal/junctional (Cardiac disorders) | 0 | 1 | 0
Constitutional Symptoms-Other (General disorders) | 1 | 1 | 0
Cardiac troponin I (cTnI) (Investigations) | 0 | 1 | 0
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PBSCC or Induction/PBSCC (N=92) | Autologous Transplants (N=65) | Dex/Thal (N=12)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 20 | 0
Hemoglobin (Blood and lymphatic system disorders) | 43 | 48 | 6
Lymphatics-Other (Blood and lymphatic system disorders) | 5 | 8 | 0
Cardiac Arrhythmia-Other (Cardiac disorders) | 1 | 12 | 0
Cardiac General-Other (Cardiac disorders) | 5 | 7 | 0
Auditory/Ear-Other (Ear and labyrinth disorders) | 1 | 0 | 1
Cushingoid appearance (Endocrine disorders) | 2 | 0 | 1
Dry eye syndrome (Eye disorders) | 0 | 2 | 1
Ocular/Visual-Other (Eye disorders) | 2 | 2 | 1
Vision-blurred vision (Eye disorders) | 2 | 4 | 2
Constipation (Gastrointestinal disorders) | 20 | 13 | 3
Diarrhea (Gastrointestinal disorders) | 13 | 41 | 1
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 6 | 0
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2 | 11 | 0
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 | 4 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 4 | 0
Heartburn/dyspepsia (Gastrointestinal disorders) | 4 | 6 | 1
Hemorrhage, GI - Lower GI NOS (Gastrointestinal disorders) | 0 | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 5 | 0
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 2 | 13 | 0
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 0 | 4 | 0
Nausea (Gastrointestinal disorders) | 28 | 44 | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 5 | 9 | 0
Vomiting (Gastrointestinal disorders) | 18 | 29 | 0
Edema: limb (General disorders) | 22 | 19 | 2
Extremity-lower (gait/walking) (General disorders) | 3 | 1 | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 41 | 41 | 7
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 5 | 20 | 0
Pain-Other (General disorders) | 2 | 2 | 1
Rigors/chills (General disorders) | 2 | 7 | 0
Allergic reaction/hypersensitivity (Immune system disorders) | 0 | 4 | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Blood (Infections and infestations) | 1 | 5 | 0
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 1 | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 0 | 4 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Catheter (Infections and infestations) | 1 | 4 | 0
Inf w/normal ANC or Gr 1-2 neutrophils - Up airway (Infections and infestations) | 3 | 3 | 3
Inf w/unknown ANC - Middle ear (otitis media) (Infections and infestations) | 0 | 0 | 1
Bruising (in absence of Gr 3-4 thrombocytopenia) (Injury, poisoning and procedural complications) | 2 | 7 | 0
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 7 | 14 | 0
AST, SGOT (Investigations) | 6 | 16 | 1
Alkaline phosphatase (Investigations) | 23 | 23 | 0
Bilirubin (hyperbilirubinemia) (Investigations) | 4 | 10 | 1
Cholesterol, serum-high (hypercholesterolemia) (Investigations) | 0 | 5 | 0
Creatinine (Investigations) | 21 | 30 | 5
GGT (gamma-glutamyl transpeptidase) (Investigations) | 1 | 10 | 0
INR (of prothrombin time) (Investigations) | 2 | 3 | 1
Leukocytes (total WBC) (Investigations) | 18 | 47 | 5
Lymphopenia (Investigations) | 9 | 11 | 2
Metabolic/Laboratory-Other (Investigations) | 4 | 5 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 10 | 46 | 3
PTT (Partial thromboplastin time) (Investigations) | 1 | 5 | 0
Platelets (Investigations) | 43 | 49 | 3
Weight gain (Investigations) | 6 | 3 | 2
Weight loss (Investigations) | 1 | 13 | 0
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 24 | 32 | 1
Anorexia (Metabolism and nutrition disorders) | 17 | 24 | 1
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 3 | 5 | 0
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 16 | 31 | 2
Dehydration (Metabolism and nutrition disorders) | 4 | 9 | 0
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 33 | 33 | 6
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 | 5 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 8 | 9 | 0
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 5 | 11 | 1
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 4 | 9 | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 18 | 15 | 0
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 10 | 18 | 1
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 2 | 4 | 0
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 9 | 14 | 0
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 7 | 4 | 0
Muscle weakness, not d/t neuropathy - Trunk (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 7 | 5 | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 6 | 5 | 2
Pain - Bone (Musculoskeletal and connective tissue disorders) | 26 | 9 | 1
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Pain - Joint (Musculoskeletal and connective tissue disorders) | 3 | 6 | 2
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 14 | 12 | 1
Dizziness (Nervous system disorders) | 13 | 17 | 3
Neuropathy: sensory (Nervous system disorders) | 14 | 8 | 5
Ocular/Visual-Other (Nervous system disorders) | 2 | 2 | 1
Pain - Head/headache (Nervous system disorders) | 11 | 14 | 1
Taste alteration (dysgeusia) (Nervous system disorders) | 2 | 15 | 0
Confusion (Psychiatric disorders) | 2 | 5 | 0
Insomnia (Psychiatric disorders) | 9 | 16 | 0
Mood alteration - depression (Psychiatric disorders) | 1 | 4 | 0
Hemorrhage, GU - Urinary NOS (Renal and urinary disorders) | 3 | 1 | 1
Proteinuria (Renal and urinary disorders) | 1 | 6 | 0
Renal failure (Renal and urinary disorders) | 9 | 9 | 0
Urinary frequency/urgency (Renal and urinary disorders) | 3 | 9 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 15 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 20 | 17 | 3
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 0
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 5 | 8 | 0
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 6 | 0
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3 | 31 | 0
Petechiae/purpura (hemorrhage into skin or mucosa) (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 6 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 8 | 19 | 2
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2 | 3 | 1
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Flushing (Vascular disorders) | 2 | 4 | 0
Hematoma (Vascular disorders) | 0 | 4 | 0
Hemorrhage/Bleeding-Other (Vascular disorders) | 10 | 5 | 0
Hypertension (Vascular disorders) | 4 | 7 | 0
Hypotension (Vascular disorders) | 15 | 21 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 4 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less